CLINICAL TRIAL: NCT07137663
Title: Investigation of the Use of Menstrual Cups in the Menstrual Health and Hygiene Management of Women Using Wheelchairs
Brief Title: The Use of Menstrual Cups in the Menstrual Health and Hygiene Management of Women Who Use Wheelchairs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hülya ULAŞLI KABAN (Other)
Responsible Party: Sponsor-Investigator, Hülya ULAŞLI KABAN, Doctoral student, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/343
Record Dates: First submitted 2025-07-25; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Menstrual Cup; Menstrual Hygiene Management; Disabled People
Keywords: Menstrual Cup; Menstrual Hygiene Management; Persons with Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Mentrual Cup Group) (Experimental): This is a single-arm study. All participants will receive a structured educational session on menstrual cup use, including hygiene, insertion and removal techniques, maintenance, and troubleshooting. Following the training, each participant will be provided with one menstrual cup for personal use. Participants will be instructed to use the cup over the course of six consecutive menstrual cycles. User satisfaction and experiences with the menstrual cup will be monitored and assessed through follow-up questionnaires at regular intervals throughout the study period. There is no control or comparator arm in this study.The study, which was semi-experimental in nature, used a repeated measures design (within-subjects design). In this type of experimental design, the participants included in the study participate in all experimental conditions. Therefore, the participants form their own control group, which increases the sensitivity of the experiment. The difference between the measurements
  Interventions: Other: Educational and practical intervention on menstrual cup use

INTERVENTIONS:
Other: Educational and practical intervention on menstrual cup use — The intervention implemented in this study is a unique approach tailored to menstrual hygiene management among women who use wheelchairs. What distinguishes this intervention from others is the combination of both education and practical support for menstrual cup use. While menstrual hygiene management in the literature generally targets the general population, this study specifically addresses the unique needs and challenges faced by women with disabilities by providing individualized menstrual cup selection and usage guidance. Additionally, the intervention includes repeated follow-ups over six menstrual cycles, allowing continuous support and monitoring of the participants' experiences. This approach aims not only to improve hygiene practices but also to enhance user satisfaction and long-term adherence. The comprehensive and personalized nature of this intervention differentiates it from most existing studies and seeks to offer practical, sustainable solutions for menstrual hygiene

SUMMARY:
This study is designed to evaluate the impact of menstrual cup use on menstrual health and hygiene management among women who use wheelchairs.In addition, the study will serve as a reference for future research that includes other groups of people with disabilities and will contribute to the literature. The main questions it aims to answer are:

How does menstrual cup use affect the menstrual hygiene management experiences of women who use wheelchairs?

What impact does menstrual cup use have on women's comfort, perception of hygiene, and participation in social life?

Do women's knowledge, attitudes, and satisfaction levels regarding menstrual cup use change over time?

Why do women who use wheelchairs choose to use or not to use menstrual cups? This quasi-experimental study will use a repeated measures design (within-subjects design). Participants included in the study will be scheduled for an appointment to receive training on menstrual cup use and to be provided with a menstrual cup. The training will be conducted face-to-face in the education room of the relevant association. During this session, the participant will first respond to the initial part of the questionnaire. Following that, she will receive training on menstrual cup use (supported by video, models, etc.), and based on the information obtained, a menstrual cup in a suitable size will be provided. The menstrual cups to be used by the participants will be supplied by the researcher.

After the initial meeting, six follow-up interviews will be conducted following the 1st, 2nd, 3rd, 4th, 5th, and 6th menstrual periods. In each session, participants will be asked to complete a follow-up-specific questionnaire, and any questions they have will be answered. Their use of the menstrual cup will be assessed during each follow-up. If a participant is not using the cup, the reasons for non-use will be explored, and if desired, the training will be repeated or individual counseling will be provided. If the participant refuses counseling or states that she no longer wishes to use the cup, she will be withdrawn from the study. If a participant drops out during the first three follow-ups, a new participant will be recruited to replace her.

ELIGIBILITY:
Inclusion Criteria:

* Having previously used a method other than a menstrual cup during menstruation,
* Being between 18 and 45 years of age,
* Having a regular menstrual cycle between 21-35 days,
* Not having a diagnosed and treated sexually transmitted infection,
* Not having a silicone allergy,
* Not having a known vaginal anatomical defect,
* Being able to actively use both arms and hands.

Exclusion Criteria:

* Planning to become pregnant,
* Having had a urogenital tract infection in the past 3 months (based on self-report),
* Having known conditions such as fibroids, endometritis, gynecological disorders, renal colic, or hydronephrosis.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2025-11-02 (Estimated); Study Completion 2027-11-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Satisfaction and Acceptability Levels in First-Time Menstrual Cup Users Who Use Wheelchairs after 6-Month Menstrual Periods Follow-Up | Baseline and 6 months.
  The study used a structured data collection form developed by the researcher based on the literature and expert opinions. The initial section (23 items) assessed participants' sociodemographic characteristics, parity, and menstrual hygiene management. Follow-up forms after menstrual periods 1-5 (18 items) evaluated menstrual cup use and menstrual hygiene management, while the final follow-up after the 6th menstrual period (23 items) included additional questions on satisfaction with menstrual cup use and perceived changes in menstrual hygiene management.
  Satisfaction with menstrual cup use was assessed using a Likert scale regarding insertion, removal, cleaning, leakage prevention, storage, odor control, comfort during daily activities, comfort during sleep, overall comfort, and perceived advantages over other menstrual hygiene products (1 = very poor, 5 = very good). Ease of use for insertion, removal, cleaning, and storage was rated as 1 = easy, 2 = not very easy, 3 = difficult.

SECONDARY OUTCOMES:
Composite questionnaires in Change from baseline in menstrual hygiene management (social life, economic aspects, and overall comfort) compared to the previous menstrual hygiene product at the 6th menstrual period. | Baseline and 6 months.
  The study used a structured data collection form developed by the researcher based on the literature and expert opinions. The initial section (23 items) assessed participants' sociodemographic characteristics, parity, and menstrual hygiene management. Follow-up forms after menstrual periods 1-5 (18 items) evaluated menstrual cup use and menstrual hygiene management, while the final follow-up after the 6th menstrual period (23 items) included additional questions on satisfaction with menstrual cup use and perceived changes in menstrual hygiene management.The menstrual periods during which participants used menstrual cups will be compared with the periods during which they used other sanitary products; perceived changes (positive/negative/no change) in economic and social life and sleep will be measured in the final follow-up form.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilbur J, Torondel B, Hameed S, Mahon T, Kuper H. Systematic review of menstrual hygiene management requirements, its barriers and strategies for disabled people. PLoS One. 2019 Feb 6;14(2):e0210974. doi: 10.1371/journal.pone.0210974. eCollection 2019. PMID 30726254
- [Background] Weerawatsopon, S., Luangdansakul, W., Prommas, S., Smanchat, B., Bhamarapravatana, K., Suwannarurk, K., 2021, Comparative study of satisfaction and acceptability between using menstrual cup versus sanitary pads in health care personnel: A randomized crossover trial, Journal of the Medical Association of Thailand, 104 (1).
- [Background] van Eijk AM, Zulaika G, Lenchner M, Mason L, Sivakami M, Nyothach E, Unger H, Laserson K, Phillips-Howard PA. Menstrual cup use, leakage, acceptability, safety, and availability: a systematic review and meta-analysis. Lancet Public Health. 2019 Aug;4(8):e376-e393. doi: 10.1016/S2468-2667(19)30111-2. Epub 2019 Jul 16. PMID 31324419
- [Background] Singh R, Agarwal M, Sinha S, Chaudhary N, Sinha HH, Anant M. Study of Adaptability and Efficacy of Menstrual Cups in Managing Menstrual Health and Hygiene: A Descriptive Longitudinal Study. Cureus. 2022 Sep 28;14(9):e29690. doi: 10.7759/cureus.29690. eCollection 2022 Sep. PMID 36187174
- [Background] Shihata, A. A., Brody, S., 2019, Five year study of a unique, eco-friendly, menstrual cup, that enhances the quality of women's lives during menstruation, Journal of Gynecology and Obstetrics, 7, 161-165.
- [Background] Rinku, N.J., 2022, Experience of female wheelchair users' personal hygiene management during menstruation. Doctoral Thesis. Bangladesh Health Professions Institute, Faculty of Medicine, the University of Dhaka, Banglades
- [Background] Hennegan J, Orozco A, Head A, Marino JL, Jayasinghe Y, Lim MSC. Menstrual cup acceptability and functionality in real-world use: A cross-sectional survey of young people in Australia. Aust N Z J Obstet Gynaecol. 2025 Jun;65(3):382-389. doi: 10.1111/ajo.13910. Epub 2024 Dec 13. PMID 39670424
- [Background] Dündar, T., Özsoy, S., 2025, The use of menstrual cups among visually impaired women, British Journal of Visual Impairment, 43 (2), 423-436.
- [Background] Dündar, T., Özsoy, S., 2020, Menstrual hijyen yönetiminde menstrual kap kullanımı, Kadın Sağlığı Hemşireliği Dergisi, 6 (1), 14-28.
- [Background] Gharacheh M, Ranjbar F, Hajinasab N, Haghani S. Acceptability and safety of the menstrual cups among Iranian women: a cross-sectional study. BMC Womens Health. 2021 Mar 13;21(1):105. doi: 10.1186/s12905-021-01259-8. PMID 33714263
- [Background] Beksinska M, Nkosi P, Zulu B, Smit J. Acceptability of the menstrual cup among students in further education institutions in KwaZulu-Natal, South Africa. Eur J Contracept Reprod Health Care. 2021 Feb;26(1):11-16. doi: 10.1080/13625187.2020.1815005. Epub 2020 Sep 17. PMID 32938248
- [Background] Averbach S, Sahin-Hodoglugil N, Musara P, Chipato T, van der Straten A. Duet for menstrual protection: a feasibility study in Zimbabwe. Contraception. 2009 Jun;79(6):463-8. doi: 10.1016/j.contraception.2008.12.002. PMID 19442783
- See also: Disability and Health Overview — https://www.cdc.gov/disability-and-health/about/index.html
- See also: Menstrual Hygiene Management — https://cdn.sida.se/publications/files/sida61960en-menstrual-hygiene-managementfeb-2016.pdf
- See also: World report on disability 2011 — https://iris.who.int/handle/10665/44575
- See also: Global report on health equity for persons with disabilities — https://www.who.int/publications/i/item/9789240063600